CLINICAL TRIAL: NCT04784104
Title: Comparison of Infraclavicular and Supraclavicular Block Approaches in Ultrasound Guided Brachial Plexus Block
Brief Title: Comparison of Infraclavicular And Supraclavicular Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Emre Şen, MD, Anesthesiology Resident, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SupraInfraTez
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia Conduction; Upper Extremity Surgery; Pain, Postoperative; Anesthesia and Analgesia; Nerve Block; Brachial Plexus Block
Keywords: Brachial plexus block; Nerve block
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Prilocaine

STUDY DESIGN:
Intervention Model Description: The study covers 2 groups. Supraclavicular block will be applied to the first group and infraclavicular block will be applied to the second group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supraclaviculer block (Experimental): The coronal oblique supraclavicular block will be applied to the first group with ultrasound guidance using a 22G 50 mm stimulator needle. 30 ml of bupivacaine (Bupivacaine HCl %0.5) and prilocaine (Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5 mcg adrenaline per ml. (14 ml. bupivacaine, 14 ml. prilocaine, 2 ml saline with 5 mcg adrenaline per ml.) Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture.
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Prilocaine HCl 2% Injectable solution; Drug: Adrenaline amp. 0.5 mg; Procedure: Ultrasound guided supraclavicular block with coronal oblique method
- Infraclaviculer block (Experimental): The lateral sagittal infraclavicular block will be applied to the second group with ultrasound guidance using a 22G 100 mm stimulator needle. 30 ml of bupivacaine (Bupivacaine HCl %0.5) and prilocaine (Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5 mcg adrenaline per ml. (14 ml. bupivacaine, 14 ml. prilocaine, 2 ml saline with 5 mcg adrenaline per ml.). Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture.
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Prilocaine HCl 2% Injectable solution; Drug: Adrenaline amp. 0.5 mg; Procedure: Ultrasound guided lateral sagittal infraclavicular block

INTERVENTIONS:
Drug: Bupivacaine HCl 0.5% Injectable Solution — 30 ml of bupivacaine (Bupivacaine HCl %0.5) and prilocaine (Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5 mcg adrenaline per ml. (14 ml. bupivacaine, 14 ml. prilocaine and 2 ml saline with 5 mcg adrenaline per ml.)
  Other Names: Bupivacaine 0.5%
Drug: Prilocaine HCl 2% Injectable solution — 30 ml of bupivacaine (Bupivacaine HCl %0.5) and prilocaine (Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5 mcg adrenaline per ml. (14 ml. bupivacaine, 14 ml. prilocaine and 2 ml saline with 5 mcg adrenaline per ml.)
  Other Names: Priloc %2
Drug: Adrenaline amp. 0.5 mg — 30 ml of bupivacaine (Bupivacaine HCl %0.5) and prilocaine (Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5 mcg adrenaline per ml. (14 ml. bupivacaine, 14 ml. prilocaine and 2 ml saline with 5 mcg adrenaline per ml.)
  Other Names: Adrenalin codex 0.5 mg 1 ml injectable solution
Procedure: Ultrasound guided supraclavicular block with coronal oblique method — The blocks will be performed by an experienced anesthesiologist with a USG guidence.
  Arms: Supraclaviculer block
Procedure: Ultrasound guided lateral sagittal infraclavicular block — The blocks will be performed by an experienced anesthesiologist with USG guidence.
  Arms: Infraclaviculer block

SUMMARY:
Ultrasound-guided brachial plexus blocks are used successfully for upper extremity surgeries. In this randomized prospective single-blind study, ASA I-II patients aged 18-65 years undergoing hand, wrist, and forearm surgery will be randomly divided into two groups. First group will receive ultrasound-guided coronal oblique supraclavicular block using a 22G, 50 mm stimulator needle, and the second group, ultrasound-guided lateral sagittal infraclavicular block using a 22G 100 mm stimulator needle. We will prepare, 30 ml of 1:1 0.5% bupivacaine and 2% prilocaine with 5 mcg adrenaline per milliliter as local anesthetic mixture. Block application time, block success, sensory and motor block levels, and postoperative analgesia time will be recorded and compared between the groups. Accordingly, the success rate of the two methods will be evaluated.

DETAILED DESCRIPTION:
In this prospective single-blind study, patients will be divided into 2 groups with the closed envelope method. Patients will be taken to the block application room before the operation. Standard monitoring (pulse oximetry, noninvasive blood pressure, ECG) will be applied to the patients. Premedication will be provided with 1mg IV midazolam after peripheral vascular access. Blocks will be performed by an experienced anesthesiologist under the guidance of USG and evaluated by another anesthesiologist who is blind to the block technique. After the antisepsis of the area, a 22G 100 mm stimulator needle will be used in the infraclavicular approach and a 22G 50 mm in the supraclavicular block. Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture. 30 ml of 1:1 0.5% bupivacaine and 2% prilocaine plus 5 mcg adrenaline per ml will be used as local anesthetic mixture. The infraclavicular block will be applied by the lateral sagittal method under USG guidance. Supraclavicular block will be applied in the coronal oblique plane while the probe is placed on the clavicle. Following the blocks, the 5th, 10th, 15th, 20th, 25th, and 30th-minute sensory block levels, 10th, 20th, and 30th-minute motor block levels will be recorded. Sensory block level; Axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain). The motor block will be evaluated with a modified bromage scale: 0: No blocks, he can lift his arm; 1: Arm is weak but active; 2: Arm is motionless but fingers are active; 3: Complete block, no movement in hand or arm.

Block success; At the 30th minute of LA application, the pinprick test will define the presence of insensibility or only a sense of touch in the musculocutaneous, radial, ulnar, median, cutaneous antebrachii nerves. If any of these nerves are not blocked, it will be considered a failed block.

Postoperative analgesia time; It will be considered as when the NRS(Numeric Rating Scale) is≥1.

Pain Score Follow-up; patients' pain scores will be recorded by checking their NRS scores at the 2nd, 6th, 12th, 24th hours.

Sensory (the time from local anesthetic injection until the patient fully perceives the upper limb) and motor (the time from local anesthetic injection until the patient's upper extremity regains full muscle strength) block time will be recorded as the block return time. Pain score during block application will be evaluated with the NRS. Block application time will be defined as the time from the moment the needle passes the skin until the local anesthetic is given and withdrawn. Block formation time will be defined as the time required to initiate anesthesia and analgesia in all 5 distal nerves. Patient and surgeon satisfaction will be evaluated as 1 = complete dissatisfaction, 2 = moderate satisfaction, 3 = full satisfaction, after the procedure. Patients will be followed up for 24 hours in terms of undesirable side effects, vascular puncture, hematoma, signs of LA toxicity, respiratory distress, pneumothorax, and horner syndrome. As rescue anesthesia, sedoanalgesia will be tried with remifentanil infusion, if it is not successful, general anesthesia will be started with a laryngeal mask. As postoperative analgesic regimen, patients will receive 3 x 1000 mg IV acetaminophen. As rescue analgesia, Tramadol 1 mg/kg IV will be ordered to be administered when the patient's NRS is 3 or more. The first time when the patient receives rescue analgesia and the total dose of rescue analgesia for the first 24 hours will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA I-II
* Patients scheduled for hand, wrist, and forearm surgery

Exclusion Criteria:

* Uncoordinated patients
* Having a disease that prevents sensory block evaluation,
* Have coagulopathy,
* Known allergies to drugs to be used,
* Those with anatomical disorders at the application points
* Pregnant patients,
* Patients under 18 years of age,
* Patients with known local anesthetic allergy,
* Patients diagnosed with sepsis and bacteriemia,
* Skin infection at the injection site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Block Formation Time | 30th minute pre-operatively
  Block formation time will be defined as the time required to initiate anesthesia and analgesia in all 5 distal nerves.
Block Application Time | During Block Application
  Block application time will be defined as the time from the moment the needle passes the skin until the local anesthetic is given and withdrawn.
Block success | At the 30th minute of LA application
  Block success; at the 30th minute of local anesthesic application, the pinprick test will define the presence of insensibility or only a sense of touch in the musculocutaneous, radial, ulnar, median, cutaneous antebrachii nerves. If any of these nerves are not blocked, it will be considered a failed block.
Sensory Block Level 5th minute | 5th minute
  Sensory block level; axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain).
Sensory Block Level 10th minute | 10th minute
  Sensory block level; axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain).
Sensory Block Level 15th minute | 15th minute
  Sensory block level; axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain).
Sensory Block Level 20th minute | 20th minute
  Sensory block level; axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain).
Sensory Block Level 25th minute | 25th minute
  Sensory block level; axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain).
Sensory Block Level 30th minute | 30th minute
  Sensory block level; axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia, and cutaneous antebrachii medialis nerve level will be evaluated with the pinprick test and its level will be recorded. (0 = painful, no block; 1 = partial block-analgesia, only tactile sensation; 2 = complete block, no pain).

SECONDARY OUTCOMES:
The Motor Block Level 10th minute | 10th minute
  The motor block will be evaluated with a Modified Bromage Scale. ( 0: No blocks, he can lift his arm; 1: Arm is weak but active; 2: Arm is motionless but fingers are active; 3: Complete block, no movement in hand or arm. )
Postoperative Analgesia Time | 24 hours post-operatively
  Postoperative analgesia time; It will be considered as when the NRS (Numeric Rating Scale) is≥1.
Pain Score Follow-up 2nd Hour | 2nd hour
  Pain Score Follow-up; patients' pain scores will be recorded by checking their NRS (Numeric Rating Scale) scores at the 2nd hour.
Block Return Time | 24 hours postoperatively
  Sensory (the time from local anaesthetic injection until the patient fully perceives the upper limb) and motor (the time from local anaesthetic injection until the patient's upper extremity regains full muscle strength) block time will be recorded as the block return time.
Patient and Surgeon Satisfaction | Immediately after the surgery
  Patient and surgeon satisfaction will be evaluated as 1 = complete dissatisfaction, 2 = moderate dissatisfaction, 3 = moderate satisfaction 4 =full satisfaction, after the procedure.
Undesirable Side Effects | 24 hours postoperatively
  Patients will be followed up for 24 hours in terms of undesirable side effects, vascular puncture, hematoma, signs of LA toxicity, respiratory distress, pneumothorax, and horner syndrome.
The Rescue Analgesia | 24 hours postoperatively
  As rescue analgesia, Tramadol 1 mg/kg IV will be ordered to be administered when the patient's NRS is 3 or more. The first time when the patient receives rescue analgesia will be recorded.
24-Hour Total Opioid Consumption | 24 hours postoperatively
  The total dose of rescue analgesia (Tramadol ) for the first 24 hours will be recorded.
Pain Score Follow-up 6th Hour | 6th Hour
  Pain Score Follow-up; patients' pain scores will be recorded by checking their NRS (Numeric Rating Scale) scores at the 6th hour.
Pain Score Follow-up 12th Hour | 12th Hour
  Pain Score Follow-up; patients' pain scores will be recorded by checking their NRS (Numeric Rating Scale) scores at the 12th hour.
Pain Score Follow-up 24th Hour | 24th Hour
  Pain Score Follow-up; patients' pain scores will be recorded by checking their NRS (Numeric Rating Scale) scores at the 24th hour.
The Motor Block Level 20th minute | 20th minute
  The motor block will be evaluated with a Modified Bromage Scale. ( 0: No blocks, he can lift his arm; 1: Arm is weak but active; 2: Arm is motionless but fingers are active; 3: Complete block, no movement in hand or arm. )
The Motor Block Level 30th minute | 30th minute
  The motor block will be evaluated with a Modified Bromage Scale. ( 0: No blocks, he can lift his arm; 1: Arm is weak but active; 2: Arm is motionless but fingers are active; 3: Complete block, no movement in hand or arm. )

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet E Şen, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Zeki T Tekgül, Assoc Prof, Study Chair — Izmir Bozyaka Training and Research Hospital; Taşkın Altay, Assoc Prof, Study Chair — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Karabağlar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurkan Y, Hosten T, Tekin M, Acar S, Solak M, Toker K. [Comparison of ultrasound-guided supraclavicular and infraclavicular approaches for brachial plexus blockade]. Agri. 2012;24(4):159-64. doi: 10.5505/agri.2012.38247. Turkish. PMID 23364778
- [Background] Grape S, Pawa A, Weber E, Albrecht E. Retroclavicular vs supraclavicular brachial plexus block for distal upper limb surgery: a randomised, controlled, single-blinded trial. Br J Anaesth. 2019 Apr;122(4):518-524. doi: 10.1016/j.bja.2018.12.022. Epub 2019 Jan 31. PMID 30857608
- [Background] Arcand G, Williams SR, Chouinard P, Boudreault D, Harris P, Ruel M, Girard F. Ultrasound-guided infraclavicular versus supraclavicular block. Anesth Analg. 2005 Sep;101(3):886-890. doi: 10.1213/01.ANE.0000159168.69934.CC. PMID 16116009